CLINICAL TRIAL: NCT02852200
Title: Screening for Frailty in Elderly Subjects Living at Home : Validation of the Modified Short Emergency Geriatric Assessment (SEGAm) Instrument
Brief Title: Screening for Frailty at Home
Acronym: SEGAm
Status: Terminated | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PO12146
Record Dates: First submitted 2016-06-17; First posted 2016-08-02 (Estimated); Last update posted 2017-10-17 (Actual); Status verified 2017-10

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other

GROUPS / COHORTS (1):
- SEGAm: Elderly community-dwelling people
  Interventions: Other: SEGAm

INTERVENTIONS:
Other: SEGAm

SUMMARY:
"Many tools to evaluate frailty have been developed. However, at the time our study was designed, none of these instruments had been validated in terms of psychometric properties. The aim of this study was to validate the modified version of the Short Emergency Geriatric Assessment (SEGAm) frailty instrument in elderly people living at home.

It was an observational, longitudinal, prospective, multicentre study, set up in four departments (Ardennes, Marne, Meurthe-et-Moselle, Meuse) in two French regions (Champagne-Ardenne and Lorraine). Subjects was aged 65 years or more, living at home, and was able to read and understand French, with a degree of autonomy corresponding to groups 5, or 6 in the AGGIR autonomy evaluation scale. Assessment included demographic characteristics, comprehensive geriatric assessment, and the SEGAm instrument. Psychometric validation was used to study feasibility and acceptability, internal structure validity, reliability, and discriminant validity of the SEGAm instrument. "

DETAILED DESCRIPTION:
Many tools to evaluate frailty have been developed. However, most are designed for use in the hospital setting, with the resultant drawback that they are not suitable for routine use in the community setting. A few tools have been developed for use in community-dwelling subjects, such as the Cardiovascular Health Study (CHS) developed by Fried from a cohort of subjects aged 65 and older; the Study of Osteoporotic Fractures (SOF); or the SHARE frailty instrument, developed in a cohort of the same name comprising subjects aged 50 years and older living at home. However, at the time our study was designed, none of these instruments had been validated in terms of psychometric properties. The aim of this study was to validate the modified version of the Short Emergency Geriatric Assessment (SEGAm) frailty instrument in elderly people living at home. It was an observational, longitudinal, prospective, multicentre study, set up in four departments (Ardennes, Marne, Meurthe-et-Moselle, Meuse) in two French regions (Champagne-Ardenne and Lorraine). Subjects was aged 65 years or more, living at home, and was able to read and understand French, with a degree of autonomy corresponding to groups 5, or 6 in the AGGIR autonomy evaluation scale. Assessment included demographic characteristics, comprehensive geriatric assessment, and the SEGAm instrument. Psychometric validation was used to study feasibility and acceptability, internal structure validity, reliability, and discriminant validity of the SEGAm instrument.

ELIGIBILITY:
Inclusion Criteria:

* Age: 65 years or more
* Living at home
* Able to read and understand French
* With a degree of autonomy corresponding to groups 5, or 6 in the AGGIR autonomy evaluation scale

Exclusion Criteria:

-

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Elderly community-dwelling people aged 65 years or over
Sampling Method: Non-Probability Sample
Enrollment: 167 (Actual)
Dates: Start 2012-06; Primary Completion 2012-07 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
The psychometric properties of SEGAm measured by questionnaire | 12 months after inclusion
  The SEGAm to be validated comprises Sheet A, which evaluates frailty per se on a 13-item scale, with each item graded either 0 (most favourable state), 1, or 2 (least favourable state), thus making it possible to classify subjects into three groups: not very frail (score ≤8), frail (8<score ≤11), and very frail (score> 11). The SEGAm was administered by social workers, ergotherapists, nurses and non-medical personnel trained in administration of the instrument.

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Reims, Reims, France

REFERENCES:
- [Background] Oubaya N, Mahmoudi R, Jolly D, Zulfiqar AA, Quignard E, Cunin C, Nazeyrollas P, Novella JL, Drame M. Screening for frailty in elderly subjects living at home: validation of the Modified Short Emergency Geriatric Assessment (SEGAm) instrument. J Nutr Health Aging. 2014;18(8):757-64. doi: 10.1007/s12603-014-0541-1. PMID 25286456